CLINICAL TRIAL: NCT01065831
Title: Faith-based Approaches in the Treatment of Hypertension (FAITH)
Acronym: FAITH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Gbenga Ogedegbe, Professor of Population Health and Medicine, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAITH 09-0558; 1R01HL092860-01A1 (NIH)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Hypertension
Keywords: motivational interviewing, lay health advisers
MeSH Terms: conditions — Hypertension | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): This MINT-TLC group will be asked to attend 12 weekly counseling meetings focused on weight loss (if overweight), limiting sodium, regular physical activity, and eating a low-fat diet that is rich in fruit and vegetables. MINT-TLC will be conducted by trained Lay Health Advisors. Participants will attend weekly group classes targeted at lifestyle changes for the first 12 weeks (intensive phase); followed by three individual MINT sessions conducted monthly for the following three months (maintenance phase). The MINT-TLC sessions aim to help participants make useful therapeutic lifestyle changes (TLC) and develop skills to maintain these changes long-term.
  Interventions: Behavioral: Motivational interviewing (MINT-TLC)
- Health Education Control Condition (Placebo Comparator): Participants randomized to this control condition will receive traditional, group health education classes for 12 weeks delivered by experts on various health topics unrelated to hypertension such as cancer, health insurance, and depression.
  Interventions: Behavioral: Motivational interviewing (MINT-TLC)

INTERVENTIONS:
Behavioral: Motivational interviewing (MINT-TLC) — The MINT-TLC lifestyle intervention lead by lay health advisers will be compared to the health education attention control condition (CC). Twenty churches will participate in the study and each church will be randomly assigned to receive either MINT-TLC or CC. They will be compared on blood pressure reduction, physical activity levels, intake of fruits and vegetables, and weight reduction.
  Other Names: Church-based lifestyle intervention; FAITH

SUMMARY:
The purpose of this study is to test the effect of a church-based lifestyle intervention on blood pressure reduction in 400 hypertensive blacks (BP> 140/90 mm hg).

DETAILED DESCRIPTION:
This study will test the effectiveness of a church-based lifestyle intervention in improving blood pressure control among 400 hypertensive blacks in a group randomized controlled trial. The lifestyle intervention will be delivered by trained lay health advisers through group-based behavioral counseling and motivational interviewing (MINT-TLC) in 24 predominantly black churches in New York City.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of hypertension
* Self-identified Black or African American
* SBP > 140 mmHg or DBP > 90 mmHg (based on the average of 3 blood pressure readings); or average SBP > 130 mm Hg or DBP > 80 mm hg (for those with diabetes or kidney disease) at the screening/baseline visits
* Able to speak English

Exclusion Criteria:

* Unable to comply with the study protocol (either self-selected or by indicating during screening that s/he could not complete all requested tasks).
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2010-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Within-individual change in systolic blood pressure and diastolic blood pressure | 6 months

SECONDARY OUTCOMES:
Levels of physical activity | 6 months
Percent change in weight | 6 months
Dietary intake of fruits and vegetables | 6 months
Proportion of blood pressure control | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Gbenga Ogedegbe, MD, Principal Investigator — NYU School of Medicine; Kristie Lancaster, PhD, Principal Investigator — NYU Steinhardt School; Antoinette Schoenthaler, EdD, Study Director — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Schoenthaler AM, Lancaster KJ, Chaplin W, Butler M, Forsyth J, Ogedegbe G. Cluster Randomized Clinical Trial of FAITH (Faith-Based Approaches in the Treatment of Hypertension) in Blacks. Circ Cardiovasc Qual Outcomes. 2018 Oct;11(10):e004691. doi: 10.1161/CIRCOUTCOMES.118.004691. PMID 30354579
- [Derived] Lancaster KJ, Schoenthaler AM, Midberry SA, Watts SO, Nulty MR, Cole HV, Ige E, Chaplin W, Ogedegbe G. Rationale and design of Faith-based Approaches in the Treatment of Hypertension (FAITH), a lifestyle intervention targeting blood pressure control among black church members. Am Heart J. 2014 Mar;167(3):301-7. doi: 10.1016/j.ahj.2013.10.026. Epub 2013 Nov 6. PMID 24576512